CLINICAL TRIAL: NCT03662880
Title: Detection of Left Atrial Thrombus by Cardiac Magnetic Resonance in Patients Undergoing Percutaneous Mitral Commissurotomy
Brief Title: Uses of CMR in Detection of Left Atrial Thrombus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Nasser Badr Hamdan, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C.M.R
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Left Atrial Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac Magnetic Resonance &Trans-esophageal echo (Other): patients undergo Percutaneous Mitral Commissurotomy will do cardiac magnetic resonance and trans esophageal echo for detection of left atrial thrombus
  Interventions: Radiation: Cardiac Magnetic Resonance; Radiation: Trans-esophageal echo

INTERVENTIONS:
Radiation: Cardiac Magnetic Resonance — Imaging modality used to detection thrombus in left atrium
Radiation: Trans-esophageal echo — a procedure in which the ultrasound probe is inserted into the esophagus and ultrasonographic images are obtained of the heart using echo and color Doppler images.

SUMMARY:
The incidence of rheumatic heart diseases have not declined in our population .Rheumatic heart diseases, often neglected by media and policy makers, is a major burden in developing countries where it causes most of the cardiovascular morbidity and mortality in young people, leading to about 250000 deaths per year worldwide. Mitralstenosis is one of the most common complications of rheumatic heart diseases in our community. A treatment of choice in suitable cases is percutaneous Mitral Commissurotomy .Preoperative evaluation for Percutaneous Mitral Commissurotomy typically requires trans-esophageal echocardiogram (TEE) for the presence of LA thrombus. TEE is currently considered the gold standard for LA thrombus detection given its favorable sensitivity and specificity . With recent advances,CMRis now becoming another reliable diagnostic method for evaluation of thrombus in the left atrium, particularly when delayed imaging is performed.

Whereas TEE is a semi-invasive procedure, CMRis totally non-invasive . Effectiveness of left ventricular thrombus detection by CMR has been validated, and it is now becoming a preferred imaging modality for evaluation of left ventricular thrombus . Moreover, in patients undergoing pulmonary vein isolation,Cardiac Magnetic Resonance was validated against TEE for LA & left atrial appendage . To our knowledge, there are few data regarding the utility of Cardiac Magnetic Resonance for detection of LA thrombus in patients undergoing Percutaneous Mitral Commissurotomy.

DETAILED DESCRIPTION:
Patients with Mitral stenosis that admitted in Assiut University hospital -Cardiovascular Department for doing Percutaneous Mitral Commissurotomy Will undergo Trans-esophageal echo and Cardiac Magnetic Resonance for detection of left atrial Thrombus and left atrial appendage thrombus. Investigators will compare the result of Cardiac Magnetic Resonance with the results of Trans-esophageal echo for seen the sensitivity and specificity of Cardiac Magnetic Resonance in compare to Trans-esophageal echo who is the gold standard imaging for detection of left atrial and left atrial appendage Thrombus.Data will be presented as mean ± standard deviation for continuous variables and frequency for categorical variables.

* Patients with and without thrombus will be compared using independent (unpaired) Student t test for continuous variables and the Fisher exact test for categorical variables, or their non-parametric equivalents, after testing the data for normality.
* Diagnostic performance of each CMR component will be calculated in the standard manner.

ELIGIBILITY:
Inclusion Criteria:

* Severe mitral stenosis .
* Significant dyspnea.
* Favorable anatomical characteristics for Percutaneous Mitral Commissurotomy as assessed by trans-thoracic echo.

Exclusion criteria:

* Critically ill patients including hemo-dynamically unstable patient.
* Implanted pacemakers/cardiac defibrillators and other electronic implants.
* Cerebral aneurysm clips.
* Pregnancy.
* Significant renal impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity of Cardiac Magnetic Resonance against Trans-esophageal echo | 24 hours
  true positive rate or probability of detection and true negative rate

SECONDARY OUTCOMES:
positive & negative predictive values, accuracy of Cardiac Magnetic Resonance against Trans-esophageal echo | 4 months
  - Positive predictive value is the probability that subjects with a positive screening test truly have the disease. Negative predictive value is the probability that subjects with a negative screening test truly don't have the disease

CONTACTS AND LOCATIONS:
Overall Officials: Amr Elbadry, MD, Principal Investigator — assiut medical school
Locations (1):
- Assiut medical school, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No